CLINICAL TRIAL: NCT05805462
Title: European microCirculatory Resistance and Absolute Flow Team: The Euro-CRAFT Registry
Brief Title: The Euro-CRAFT Registry
Acronym: Euro-CRAFT
Status: Active, not recruiting | Type: Observational
Sponsor: CoreAalst BV (Industry)
Collaborators: Hexacath, France (Industry)
Responsible Party: Sponsor
Other Study IDs: CRI-080
Record Dates: First submitted 2023-03-02; First posted 2023-04-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Coronary Microvascular Disease
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Euro-CRAFT Registry is a prospective, multicentric, international registry of patients undergoing functional assessment of the coronary microcirculation using the continuous thermodilution technique. Angina and quality of life questionnaires (Seattle Angina Questionnaire 19 - SAQ19, ORBITA app) will be obtained at baseline, at 6 months, and 1-year follow-up. Clinical follow-up will be performed at 1 year (optionally until 5 years).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Stable patients should have complaints of chest pain suspected of angina pectoris or other symptoms raising the suspicion of IHD and non-obstructive epicardial coronary arteries on invasive coronary angiography (ICA, diameter stenosis of less than 50%) with an FFR >0.80.
* Any other clinical scenario (including in the context of ACS) prompting the physician to assess the function of the coronary microvasculature.

Exclusion Criteria:

* Unable to provide consent
* Unstable hemodynamics
* Ongoing chest pain.
* Previous CABG
* Moderate to severe valvular heart disease
* Uncontrolled or recurrent ventricular tachycardia.
* Active liver disease or hepatic dysfunction, defined as AST or ALT > 3 times the ULN.
* Comorbidity with life expectancy <= 2 years.
* Severe renal dysfunction, defined as an eGFR <30 mL/min/1.73 m2.
* Subject is currently participating in another investigational drug or device clinical study.
* Presence of other anatomic or comorbid conditions, or other medical, social or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients in whom physiological assessment of the microcirculatory function including continuous coronary thermodilution has been performed with a Pressure-wire X within the context of routine clinical care.
Sampling Method: Probability Sample
Enrollment: 671 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2030-09-22 (Estimated)

PRIMARY OUTCOMES:
The rate of MACCE between patients with and without CMD based on MRR at 1-year follow-up. | 12 months follow-up
  Rate of Major Adverse Cardiac and Cerebrovascular Events at one year (MACCE defined as cardiovascular death, angina and heart failure related hospitalisations and stroke) between patients with and without Coronary Microvascular Disease (CMD) defined according to thermodilution derived metrics (Microvascular Resistance Reserve, MRR).

SECONDARY OUTCOMES:
Relationship between MACCE's and each thermodilution- derived metrics of microvascular function | 12 months follow-up
  Relationship between Major Adverse Cardiac and Cerebrovascular Events (MACCE defined as cardiovascular death, angina and heart failure related hospitalisations and stroke) and each thermodilution-derived metrics of microvascular function (i.e. absolute hyperemic flow, absolute hyperemic resistance, Index of Microvascular Resistance, and Coronary Flow Reserve)
Relationship between the presence and severity of angina, assessed by SAQ- 19, and each individual thermodilution-derived metrics of microvascular function | 12 months follow-up
  Relationship between the presence and severity of angina, assessed by Seattle Angina Questionnaire 19, and each individual thermodilution-derived metrics of microvascular function (i.e., absolute hyperemic flow, absolute hyperemic resistance,Index of Microvascular Resistance and Coronary Flow Reserve).
Relationship between the presence and severity of angina, assessed by the ORIBTA Euro-CRAFT app, and each individual thermodilution-derived metrics of microvascular function | 12 months follow-up
  Relationship between the presence and severity of angina, assessed by the ORBITA Euro-CRAFT app, and each individual thermodilution-derived metrics of microvascular function (i.e., absolute hyperemic flow, absolute hyperemic resistance, Index of Microvascular Resistance and Coronary Flow Reserve).
Safety of continuous and bolus thermodilution measurements, as assessed by adverse event registration. | 12 months follow-up
  Safety of continuous and bolus thermodilution measurements, as assessed by adverse event registration.
To determine cut-off values of thermodilution-derived indices | 12 months follow-up
  To determine cut-off values of thermodilution-derived indices (i.e. absolute hyperemic flow, absolute hyperemic resistance, Index of Microvascular Resistance and Coronary Flow Reserve to assess the presence of Coronary Microvascular Disease.
To assess the prevalence of Coronary Microvascular Disease based on Microvascular Resistance Reserve in patients with angina and non-obstructive coronary artery disease (NOCAD) | 12 months follow-up
  To assess the prevalence of CMD based onMicrovascular Resistance Reserve (MRR) in patients with angina and non-obstructive coronary artery disease (NOCAD)

CONTACTS AND LOCATIONS:
Locations (19):
- OLV Ziekenhuis Aalst, Aalst, Belgium
- Righospitalet, Copenhagen, Denmark
- University of Mainz, Mainz, Germany
- Netherlands (3):
  - Catharina Hospital, Eindhoven
  - Radboud Hospital, Nijmegen
  - Maasstad Ziekenhuis, Rotterdam
- University Clinical Center of Serbia, University of Belgrade, Belgrade, Serbia
- Spain (3):
  - University Hospital Puerta del Mar, Cadiz
  - Clinica La Princesa, Madrid
  - San Carlos Hospital, Madrid
- University Hospital Lausanne, Lausanne, Switzerland
- United Kingdom (8):
  - Royal United Hospital Bath NHS Foundation Trust, Bath
  - Bristol Heart Institute, Bristol
  - Basildon Hospital, Essex
  - Golden Jubilee National Hospital, Glasgow
  - Imperial College, London
  - Royal Brompton Hospital, London
  - St. Thomas Hospital, King's College, London
  - Oxford University Hospitals, Oxford

IPD SHARING:
Plan to Share IPD: No